CLINICAL TRIAL: NCT01621932
Title: Anterior Capsulectomy vs. Repair in Direct Anterior THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101105A
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Total Hip Arthroplasty
Keywords: Anterior approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical approach 1 (Active Comparator): Direct anterior surgical approach with capsulectomy
  Interventions: Procedure: Direct anterior approach with capsulectomy
- Surgical approach 2 (Active Comparator): Direct anterior approach without capsulectomy
  Interventions: Procedure: Direct anterior approach without capsulectomy

INTERVENTIONS:
Procedure: Direct anterior approach with capsulectomy — Direct anterior approach with capsulectomy
  Arms: Surgical approach 1
Procedure: Direct anterior approach without capsulectomy — Direct anterior approach without capsulectomy
  Arms: Surgical approach 2

SUMMARY:
Randomized prospective study comparing the anterior capsule repair vs capsulectomy with regards to post-operative pain and range of motion outcomes in elective primary unilateral direct anterior approach THA for osteoarthritis. Visual Analog Scores (VAS) will be recorded for preoperative and postoperative months 1 and 4. Hip range of motion will be assessed by goniometer measurements and lateral hip radiographs in maximum flexion.

The purpose of the study is to compare post-operative pain control and hip range of motion between two surgical techniques (anterior capsular repair vs. anterior capsulectomy) during direct anterior total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral primary total hip arthroplasty Direct anterior surgical approach Osteoarthritis diagnosis 18 years of age or older

Exclusion Criteria:

* Bilateral primary total hip arthroplasty Revision hip arthroplasty Avascular necrosis of the hip Rheumatoid arthritis of the hip Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Hip flexion | postoperative 4 months

SECONDARY OUTCOMES:
Visual analog scale-pain | 4 months and 12 months post operative

CONTACTS AND LOCATIONS:
Overall Officials: John Masonis, MD, Principal Investigator — OrthoCarolina, P.A.
Locations (1):
- OrthoCarolina, P.A., Charlotte, North Carolina, United States